CLINICAL TRIAL: NCT02491788
Title: Examination of the Effectiveness of Suvorexant in Improving Daytime Sleep in Shift Workers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry); Stanford University (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Associate Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-34778
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Sleep Disorder, Shift-Work
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Experimental): 10 mg of suvorexant 30 minutes prior to daytime sleep opportunity
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Placebo pill 30 minutes prior to daytime sleep opportunity
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant
  Other Names: Belsomra
  Arms: Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that ingestion of the wake-inhibiting drug suvorexant 30 minutes prior to daytime sleep initiation in individuals working overnight shifts will significantly improve both objective (total sleep time, sleep efficiency, wake after sleep onset) and subjective (sleep quality) measures of daytime sleep.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 (older individuals excluded due to altered sleep-related circadian signaling)
* Males and females
* Shift worker

  * Minimum of three months of prior shift work
  * Will work minimum of four nights per week or 32 hours of night shift per week during study
  * "Night work" defined as having at least six hours of work occurring between 8 PM and 8 AM and no longer than 12 hours on shift
* Presence of DSM-5 defined Circadian Rhythm Sleep-Wake Disorder: Shift Work Type

  * Insomnia (SE < 88%) during attempted daytime sleep or excessive sleepiness during nocturnal wake

Exclusion Criteria:

* Currently or planning to become pregnant
* Currently breastfeeding
* Inadequate opportunity (<7 hours) for daytime sleep after shift work
* Use of sleep aids during the study period. Includes as needed or continuous use of prescription, non-prescription, and naturopathic pharmacotherapies
* Diagnosis or detection (during study) of sleep disordered breathing (AHI>10) on home sleep testing; referral to clinical sleep program will be offered
* Diagnosis of narcolepsy
* Restless Legs Syndrome
* >600 mg caffeine intake per night shift or use of prescription stimulant medication during night shift
* Rotational or irregular work shifts during study
* Use of digoxin for six months prior to or during study
* Use of strong (e.g., etoconazole, itraconazole, posaconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, boceprevir, telaprevir, telithromycin, conivaptan) or moderate (e.g., amprenavir, aprepitant, atazanavir, ciprofloxacin, diltiazem, erythromycin, fluconazole, fosamprenavir, grapefruit juice, imatinib, verapamil) CYP3A inhibitors or CYP3A inducers (e.g., rifampin, carbamazepine, phenytoin) for six months prior to or during study
* Severe hepatic impairment
* Unstable or severe medical or psychiatric condition

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
All relevant data will be provided in the publication

REFERENCES:
- [Derived] Zeitzer JM, Joyce DS, McBean A, Quevedo YL, Hernandez B, Holty JE. Effect of Suvorexant vs Placebo on Total Daytime Sleep Hours in Shift Workers: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206614. doi: 10.1001/jamanetworkopen.2020.6614. PMID 32484552

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: 10+ mg of suvorexant 30 minutes prior to daytime sleep opportunity
  Suvorexant
- Placebo: Placebo pill 30 minutes prior to daytime sleep opportunity
  Placebo
Period: Overall Study
Arm/Group | Drug | Placebo
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Drug: 10 mg of suvorexant 30 minutes prior to daytime sleep opportunity
  Suvorexant
- Total: Total of all reporting groups
Arm/Group | Drug | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.9) | 35.1 (9.33) | 37.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Total Sleep Time
Description: Change in average of the total amount of sleep occurring during daytime sleep episodes following night shift work, as compared to baseline
Time Frame: Daytime sleep will be examined from baseline to after 3 weeks
Measure: Mean (Standard Error); unit: hours/sleep opportunity
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 8 | 11
hours/sleep opportunity | 1.83 (0.62) | -0.33 (0.49)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 2.16, Standard Error of Mean 0.75

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Weekly and ad libitum telephone assessment with project coordinator
Arm/Group | Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=8) | Placebo (N=11)
Facial swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant felt that facial swelling occurred contemporaneously with onset of taking the study medication (placebo). Participant decided to remain in study. Unblinding was not revealed to participant or study team who assessed the data.
Fatigue (Nervous system disorders) | 0 (0) | 1 (1) — Participant felt taking the study medication (placebo) made it more difficult to run in the evening. Participant decided to remain in study. Unblinding was not revealed to participant or study team who assessed the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT02491788/Prot_SAP_001.pdf